CLINICAL TRIAL: NCT00202904
Title: A Multicenter, Randomized, Parallel Groups, Placebo-Controlled Study Comparing the Efficacy, Safety, and Tolerability of the Daily Co-Administration of Ezetimibe 10 mg or Ezetimibe Placebo to Ongoing Treatment With Atorvastatin 10 mg in Subjects With Primary Hypercholesterolemia and Coronary Heart Disease
Brief Title: Effectiveness and Safety of Ezetimibe Added to Atorvastatin in Patients With High Cholesterol and Coronary Heart Disease (Study P03740)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03740
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
Keywords: ezetimibe; atorvastatin; hypercholesterolemia; coronary heart disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: ezetimibe
- Arm 2 (Active Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10 mg tablets, one tablet taken daily with atorvastatin 10 mg daily for 6 weeks
  Other Names: Zetia, SCH 58235
  Arms: Arm 1
Drug: placebo — placebo tablets matched to ezetimibe, one tablet taken daily with atorvastatin 10 mg daily for 6 weeks
  Arms: Arm 2

SUMMARY:
This is a multicenter, randomized, parallel group, placebo controlled study designed to evaluate the efficacy, safety, and tolerability of ezetimibe added to ongoing atorvastatin therapy compared with ongoing atorvastatin treatment alone. This study will involve subjects with primary hypercholesterolemia and coronary heart disease (CHD) who are currently being treated with atorvastatin and who would benefit from additional reduction in low-density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
This multicenter, randomized, parallel groups, placebo-study is designed for subjects with primary hypercholesterolemia [plasma LDL-C concentrations between >= 2.6 mmol/L (100 mg/dL) to <= 4.1 mmol/L (160 mg/dL) and triglyceride concentrations of < 3.99 mmol/L (350 mg/dL) and coronary heart disease who are currently being treated with atorvastatin 10 mg and would benefit from additional reduction in LDL-C.

This study will assess whether the daily co-administration of ezetimibe 10 mg to ongoing treatment with atorvastatin 10 mg will be more effective than treatment with atorvastatin 10 mg alone in further reducing LDL-C concentrations and in achieving LDL-C target goal as defined by the ESC or National Cholesterol Education Program (NCEP) guidelines at the time of database lock.

The primary objective is to compare the efficacy of ezetimibe 10 mg added daily to ongoing treatment with atorvastatin 10 mg versus ezetimibe placebo added daily to ongoing treatment with atorvastatin 10 mg in reducing the concentration of LDL-C at endpoint after 6 weeks of treatment.

The secondary objective is to compare the efficacy of ezetimibe 10 mg added to ongoing treatment with atorvastatin 10 mg daily versus ezetimibe placebo added to ongoing treatment with atorvastatin 10 mg daily after 6 weeks of treatment with respect to:

* The percentage of subjects who achieve the target LDL-C goal as defined by the ESC or NCEP guidelines at the time of database lock.
* Change in the concentrations of total cholesterol, HDL-C and triglycerides.
* Safety and tolerability. Approximately 200 subjects will be enrolled into the study to insure that at least 160 subjects complete the study. Each site will enroll approximately 20 subjects for a total of approximately 200 subjects.

The duration of the study for each subject will be approximately 7 weeks. Each subject will be scheduled for 3-4 study visits. Visits 1 and 2 are screening visits; these visits may be combined. At Visit 3, those subjects who meet the enrollment criteria will be randomized to one of two treatment groups: ezetimibe 10 mg or ezetimibe placebo to be taken with ongoing open-label atorvastatin 10 mg/day. Randomization will be stratified based on the LDL-C level at Visit 3: < 3.3 mmol/L (130 mg/dL) or >= 3.3 mmol/L (130 mg/dL). Subjects will be treated for 6 weeks and then return for a final visit, Visit 4.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >=18 years and <=75 years of age.
* Subjects must have an LDL-C concentration >=2.6 mmol/L (100 mg/dL) to <=4.1 mmol/L (160 mg/dL) using the Friedewald calculation available at the time of randomization (Baseline Visit).
* Subjects must have triglyceride concentrations of <3.99 mmol/L (350 mg/dL) at Visit 3 (Baseline Visit).
* Subjects must have documented coronary heart disease (CHD). For the purposes of this study, CHD will include one or more of the following features:

  * Documented stable angina (with evidence of ischemia on exercise testing)
  * History of myocardial infarction
  * History of percutaneous coronary intervention (primarily percutaneous coronary transluminal angioplasty (PCTA) with or without stent placement)
  * Symptomatic peripheral vascular disease (claudication)
  * Documented history of unstable angina or non-Q wave myocardial infarction.
* Subject must be currently taking atorvastatin 10 mg daily and by history has taken 80% of daily doses for the preceding 6 weeks prior to Visit 3 (Baseline Visit).
* Subjects must have liver transaminases (alanine aminotransferase (ALT), aspartate aminotransferase (AST) <50% above the upper limit of normal, with no active liver disease, and creatinine kinase (CK) <50% above the upper limit of normal at Visit 3 (Baseline Visit).
* Clinical laboratory tests (complete blood count (CBC), blood chemistries, urinalysis) must be within normal limits or clinically acceptable to the investigator at Visit 3 (Baseline Visit).
* Subjects must have maintained a cholesterol lowering diet and exercise program for at least 4 weeks prior to the study and be willing to continue the same diet and exercise program during the study.
* Subjects must report a stable weight history for at least 4 weeks prior to entry into study at Visit 3 (Baseline Visit).
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, must have been maintained on a stable dose and regimen for at least 8 weeks and be willing to continue the same regimen for the duration of the study.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must be free of any clinically significant diseases other than hyperlipidemia or coronary heart disease that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and must agree to remain on their current cholesterol-lowering diet and their current exercise regimen for the duration of the study.

Exclusion Criteria:

* Subjects whose body mass index (BMI=weight [kg]/height2[m]) is >=30 kg/m2 at Visit 3 (Baseline Visit).
* Subjects who consume >14 alcoholic drinks per week. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Any condition or situation which, in the opinion of the investigator, might pose a risk to the subject or interfere with participation in the study.
* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Subjects who have the following medical conditions:

  * Congestive heart failure defined by New York Heart Association (NYHA) as Class III or IV.
  * Uncontrolled cardiac arrhythmia.
  * Myocardial infarction, acute coronary insufficiency, coronary artery bypass surgery, or angioplasty within 3 months of Visit 3 (Baseline Visit).
  * Unstable or severe peripheral artery disease within 3 months of Visit 3 (Baseline Visit).
  * Newly diagnosed or currently unstable angina pectoris.
  * Uncontrolled hypertension (treated or untreated) with systolic blood pressure >160 mmHg or diastolic >100 mmHg at Visit 3 (Baseline Visit).
  * Type I or Type II diabetes mellitus.
  * Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, i.e., secondary causes of hyperlipidemia, such as secondary hypercholesterolemia due to hypothyroidism (TSH above upper limit of normal) at Visit 3. Subjects with a history of hypothyroidism who are on a stable therapy of thyroid hormone replacement for at least 6 weeks are eligible for enrollment if thyroid-stimulating hormone (TSH) levels are within normal limits at Visit 3 (Baseline Visit).
  * Impaired renal function (creatinine > 2.0 mg/dL) or nephrotic syndrome at Visit 3 (Baseline Visit).
  * Disorders of the hematologic, digestive, or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
  * Known human immunodeficiency virus (HIV) positive.
  * Cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
  * History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Subjects who are on any of the following concomitant medications:

  * Medications that are potent inhibitors of CYP3A4, including cyclosporine, systemic itraconazole, fluconazole, and ketoconazole, erythromycin or clarithromycin, nefazodone, mibefradil, protease inhibitors and large amounts of grapefruit juice (>1 quart/day).
  * Lipid-lowering agent: niacin (>200 mg/day) and resins taken within 5 weeks, fibric acid derivatives taken within 8 weeks, and probucol taken within one year prior to Visit 3 (Baseline Visit).
  * Over the counter lipid lowering agents such as fish oils, garlic and cholestin taken within 5 weeks prior to Visit 3 (Baseline Visit).
  * Oral corticosteroids unless used as replacement therapy for pituitary/adrenal disease and the subject is on a stable regimen for at least 6 weeks prior to Visit 3 (Baseline Visit).
  * Subjects who are currently using cardiovascular medication and have not been on a stable regimen for at least 6 weeks prior to Visit 3 (Baseline Visit) and it is expected to change during the study.
  * Subjects who are currently using psyllium, other fiber-based laxatives, and/or any other over-the-counter (OTC) therapy known to affect serum lipid levels (phytosterol margarine), and have not been on a stable regimen for at least 5 weeks prior to study entry Visit 3 (Baseline Visit) and who do not agree to remain on this regimen throughout the study.
  * Subjects who are currently using orlistat or sibutramine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of ezetimibe 10 mg added daily to ongoing treatment with atorvastatin 10 mg versus placebo added daily to ongoing treatment with atorvastatin 10 mg in reducing the concentration of LDL-C at endpoint | after 6 weeks of treatment

SECONDARY OUTCOMES:
To compare the percentage of subjects who achieve target LDL-C goal (as defined by the ESC or NCEP guidelines at the time of database lock) with ezetimibe 10 mg added to atorvastatin 10 mg daily versus placebo added to atorvastatin 10 mg daily | after 6 weeks of treatment
To compare the change in concentrations of total cholesterol, HDL-C and triglycerides with ezetimibe 10 mg added to atorvastatin 10 mg daily versus placebo added to atorvastatin 10 mg daily | after 6 weeks of treatment
To compare the safety and tolerability of ezetimibe 10 mg added to atorvastatin 10 mg daily versus placebo added to atorvastatin 10 mg daily | after 6 weeks of treatment